CLINICAL TRIAL: NCT02132273
Title: Use of an Educational Story to Prepare Children With Developmental Disabilities for Overnight Polysomnography
Brief Title: Use of an Educational Story to Prepare Children With Developmental Disabilities for Sleep Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Accardo (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Sponsor-Investigator, Jennifer Accardo, Assistant Professor of Neurology, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Organization: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 100-EP-13
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Developmental Disabilities; Sleep Disorders; Polysomnography; Preparation for Medical Procedure; Child
MeSH Terms: conditions — Developmental Disabilities; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Story (Experimental): Participants receiving this intervention will have access to the educational story as they prepare for the overnight sleep study.
  Interventions: Other: Educational Story
- Typical Preparation (No Intervention): Participants will receive traditional materials, directions, what to bring list, only. They will not recieve access to educational story

INTERVENTIONS:
Other: Educational Story — Educational story with pictures illustrating overnight polysomnography procedure accompanied by simple narrative.
  Other Names: "The Sleep Study Story"
  Arms: Educational Story

SUMMARY:
The investigators hypothesize that use of an educational story with pictures illustrating overnight sleep study procedure (also called polysomnography or PSG)accompanied by simple narrative will be a cost-effective, readily accepted intervention that will contribute to successful completion of sleep studies among children with disabilities. Children who have been referred for a clinical sleep study at Kennedy Krieger Institute (KKI) will be enrolled and randomized to either recieve usual care (discussion of polysomnography with referring clinicians) or educational story intervention. Both groups of participants will be asked to complete questionnaries before and after the sleep study. Set-up for the sleep study will be videotaped so that behavior of the child can be evaluated. The investigators will evaluate whether successful study completion differs between the two groups.

DETAILED DESCRIPTION:
This pilot study is a prospective clinical trial comparing parent knowledge of, and child outcomes for clinically indicated PSG which is part of routine care. Comparisons will take place before and after either educational intervention or usual clinical care preparing children for PSG at KKI. Interested families will be recruited through the Kennedy Krieger Institute (KKI) Sleep Disorders Clinic and flyers will be distributed to other KKI subspecialty clinics in which clinically indicated PSG may be ordered. Families for whose children PSG is clinically recommended in KKI Sleep Disorders Clinic will have informed consent obtained from parents and assent from children in clinic, and randomization will occur at that time. Alternately, families for whose children PSG is clinically recommended in that clinic or others may contact the research coordinator for phone screening (telephone script attached) in order to be consented and assented; randomization will then take place once informed consent is received. Families randomized to the educational story intervention group will receive a printed copy of the educational story, as well as instructions on how to use it. Families randomized to the standard clinical care group will receive a set of pictures used in standard clinical care without an accompanying educational story.

The educational story has been developed by the Primary Investigator, who is board certified in Pediatrics and Sleep Medicine, and the Co-Investigator, who has extensive training in child clinical and pediatric psychology. It has also been reviewed by professionals at the KKI Center for Autism and Related Disorders with experience in developing educational materials for children with disabilities. There is a single version of this story that parents will be given to take home and review with their child. It is a short, upbeat narrative about a boy who comes to the investigators pediatric sleep laboratory for his first PSG. It is illustrated with color photographs depicting the entire PSG process (arrival at the laboratory, each step of PSG setup, the final appearance of the child with monitoring applied, the child asleep, and departure the following morning after a successful PSG). The text has a Flesch-Kincaid grade level of 2.5, and Flesch reading ease of 89.4.

Research procedures prior to PSG include completion of the following questionnaires:

1. Demographic questionnaire
2. Pre-PSG knowledge questionnaire
3. Pediatric Symptom Checklist
4. Parent Beliefs Scale

These questionnaires will be done 2-3 weeks prior to the night of the PSG.

All families will receive a phone call one week prior to PSG reminding them of their upcoming procedure, and for families in the intervention group, reminding them to review the social story. Parents in the intervention group will be asked to review the story at least 3 times with their child.

Research procedures for parents on arrival the night of the clinically indicated PSG include the following:

1. Post-PSG knowledge questionnaire (on arrival at the laboratory)
2. Parent Beliefs Scale (on arrival at the laboratory)

Because Dr. Paasch and Dr. Accardo are blinded to the randomization of study subjects, they will be able to score pre-PSG questionnaires and enter data as needed throughout the study.

Research procedures to be completed by sleep technicians the night of the study are the following:

1. Adapted Wong-Baker FACES distress scale (based on child distress)
2. Audio and video recording of equipment setup. Clinical PSG is accompanied by audio and video recording as part of routine care, but the investigators will extend the video recording to include equipment setup specifically for the purpose of research in order to quantify duration of setup time and number of escape behaviors.

Research procedures for parents prior to discharge from the laboratory will consist of a post-PSG qualitative questionnaire (prior to discharge from the laboratory) regarding their experience in the laboratory. In the case of the intervention group, they will also be asked how the educational story was helpful and whether parents recommended changes to make it more helpful in future.

After completion of the PSG and completion of questionnaires, the study is complete. Therefore the average length of time over which the study takes place, is approximately 3-4 weeks.

Following completion of the clinically indicated PSG performed for clinical care purposes, several steps will occur:

1. The PSG will be scored per laboratory protocol by a certified registered PSG technician.
2. The Primary Investigator, Dr. Accardo, will review data and generate a clinical interpretation of the PSG detailing whether any sleep concerns or diagnoses were identified during the study.
3. Audio and video recording will be reviewed by co-investigator Dr. Valerie Paasch based on the Pediatric Behavior Adjustment Scale (PBAS) to document any child distress and complete task analysis to document the steps which were completed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical recommendation for polysomnography to be performed at KKI Clinical Neurophysiology Laboratory
* age 4 -17 years
* adequate health to tolerate procedure without additional nursing care
* English speaking caregiver, over 18 years of age
* Caregiver must have full guardianship of child participant
* Caregiver must be able to complete written questionnaires and read the educational story to their child
* Caregiver must be able to accompany child participant to the sleep study

Exclusion Criteria:

* non-english speaking children
* children in foster care or wards of the state
* child with absence of developmental disability
* child with presence of severe-profound intellectual disability
* child with severe disruptive or aggressive behaviors
* recommended for titration study (CPAP and/or supplemental oxygen)
* children requiring behavioral desensitization prior to sleep study.
* Caregivers that are non-English Speaking
* Caregivers that are under 18 years of age
* foster parents or temporary guardians
* cargivers with inability to reach educational story and/or complete questionnaires.
* caregiver is unable to accompany the child to the sleep study

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Task Analysis and Pediatric Behavior Adjustment Scale | PSG Set-UP 2- 3 weeks after enrollment
  Task Analysis: Quantification of number of PSG steps technician was able to complete during setup
  Pediatric Behavior Adjustment Scale: Quantification of child escape behaviors during PSG equipment setup based on standardized review of audio and video recording

SECONDARY OUTCOMES:
Parent Completed Questionnaires | 2-3 weeks prior to PSG, and night of Sleep Study
  1. Demographic Questionnaire: Parent and child demographics
  2. Pre-PSG Knowledge Questionnaire: Baseline parent knowledge about PSG
  3. Pediatric Symptom Checklist: Cognitive, emotional and behavioral symptoms in child
  4. Modified PSG Parent Beliefs Scale: Parent perceptions of parent ability to help child cope with procedure as well as child ability to cope with procedure
  5. Post-PSG Knowledge Questionnaire: Post-intervention parent knowledge about PSG
  6. Post-PSG Qualitative Questionnaire: Qualitative parent feedback on child and parent PSG experience and on educational intervention if applicable

OTHER OUTCOMES:
Educational Story Questionnaire | Morning after PSG (Treatment Group Only) 3-4 weeks after enrollment.
  Evaluation pf the parent's use and beliefs regarding the effectiveness of the educational story

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Accardo, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No